CLINICAL TRIAL: NCT02657109
Title: Influence of Early Mobilization Protocol in Heart Valve Replacement on Heart Rate Variability and Oxidative Stress
Brief Title: Influence of a Rehabilitation in Valve Replacement on Heart Rate Variability and Oxidative Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Metodista de Piracicaba (Other)
Responsible Party: Principal Investigator, Rodrigo Santiago Barbosa Rocha, Phd, PHD STUDENT, Universidade Metodista de Piracicaba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 37/2014
Record Dates: First submitted 2016-01-11; First posted 2016-01-15 (Estimated); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Cardiac Valve Disease
Keywords: valve replacement; physical therapy; early mobilization
MeSH Terms: conditions — Heart Valve Diseases | interventions — Physical Therapy Modalities; Early Ambulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator): Participants are submitted to cardiac rehabilitation protocol of the hospital where it will be conducted the study, which consists in respiratory exercises of 3 series Inspirations Maximum Sustained for 10 reps, 3 sets of 20 repetitions metabolic exercises with dorsiflexion and plantar flexion and ankle and wrist extension and fingers of the upper limbs. Assessment of heart rate varibility and oxidative stress carried out before the heart valve replacement surgery , the first day of postoperative and on the fifth postoperative day
  Interventions: Other: physical therapy procedure
- Early mobilization (Active Comparator): Participants performed exercise in cycle ergometer of lower Limbs, pedaling for 20 consecutive minutes at a moderate level with Heart Rate Assessment and the Borg scale to evaluate the Voluntary Comfort. Assessment of heart rate varibility and oxidative stress carried out before the heart valve replacement surgery , the first day of oepratório post and on the fifth postoperative day
  Interventions: Other: physical therapy procedure

INTERVENTIONS:
Other: physical therapy procedure — physiotherapy exercises conducted in early way for the rehabilitation of patients in the postoperative period of cardiac valve replacement.
  Other Names: early mobilization

SUMMARY:
4 consecutive days with volunteers between the first and fourth postoperative period of cardiac valve replacement. The volunteers are randomized into 2 groups: the Control Group submitted to cardiac rehabilitation protocol of the hospital where it will be conducted the study, which consists of respiratory and metabolic exercises. The second group, called Early Mobilization Group in addition to the aforementioned exercises will be added exercise in cycle ergometer. For the implementation of rehabilitation protocol in the early mobilization group volunteers will be placed in a sitting position in the bed with the backrest raised to 45 °. The exercise in cycle ergometer will be held for 20 minutes on four consecutive days of active mode, the training load shall be such that the voluntary maintained throughout training a level of fatigue, maintaining level of heart rate predicted for age increased by 70% and 1 w / cm2 every minute to keep the parameter within the standards. The evaluation of heart rate variability with the Polar monitor RS800CX brand model before surgery was performed first postoperative day and fifth postoperative day in the control groups and early mobilization.

DETAILED DESCRIPTION:
The valve disorders are a special group of heart diseases with long period without clinical manifestations, when there is the appearance of symptoms, the patient is a likely candidate for surgery. In many surgical complications can occur, including the respiratory cause and immobility in bed culminating in the need for intensive care. Early mobilization exercises conducted by physical therapy in critically ill patients is to minimize complications related to immobility in bed from surgery that is performed in exchanges of heart valves. To investigate the influence of a cardiac rehabilitation program on cardiac function (Heart Rate Varibility) and free radicals (oxidative stress) in patients undergoing surgical heart valve replacement. The study is being conducted at the Clinical Hospital Gaspar Viana of Belém, in March 2014 period to March 2016, with the proposing institution the Methodist University of Piracicaba. The study included 60 volunteers aged 18 to 60 year old male with surgery scheduling of heart valve replacement. The volunteers were divided into 2 groups the control group who underwent rehabilitation proposed by the hospital with simple exercises like deep breathing exercises to improve cough, move your arms and rhythmically legs to maintain joint mobility, the second group It was called Early Mobilization Group, where volunteers beyond rehabilitation protocol proposed by the hospital, held exercises in a cycle ergometer, The volunteers were instructed to pedal lying comfortably with moderate intensity for 30 minutes. All groups performed this protocol lasting 4 days. Oxidative stress was analyzed and cardiac function before surgery, after surgery in the first and fifth postoperative. The Oxidative Stress is analyzed by puncturing a drop of blood and to analyze the photographed area coagulum formed. Cardiac function (Heart Rate Variability) will be analyzed using a heart rate monitor brand Polar® RS800CX model being evaluated lying down, then the data is transferred to the computer and analyzed in a program called Kubios HRV. After collecting the data will be analyzed in Biostat 5.2 program. The possible risks to the research subject is the inconvenience of collecting the blood sample, the onset of pain resulting from the mobilization of the rehabilitation protocol. However, the emergence of at least one of the risks mentioned above, the procedure and / or service must be stopped and perform passive stretching or temporary home until everything returns to normal. In addition, there may be a risk of contamination to volunteer for collecting blood, however this risk is minimized when using materials such as sterile needles and blades. The research brings benefit as increased range of motion and muscle strength, decreased pain, functional improvement, providing improvement in quality of life and functional independence and reduced hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers underwent cardiac valve replacement surgery
* Using median sternotomy
* Aged 30 60 years
* Pulse saturation greater than 90%
* BMI ranging between 18.5 and 25 kg / m2

Exclusion Criteria:

* Less than 30 years or over 60 years of age
* Other type of heart surgery than valve replacement, as well valve re-replacement
* Unconscious and level of the Glasgow Coma below scale 15
* Cardiac arrhythmias
* With electrolyte disturbances
* With pleural diseases such as pneumothorax, empyema or pleural effusion
* Circulatory failure acute
* Infections in either system
* Patients with coagulation disorders
* Pulse oxygen saturation lower than 90% even with supplementary oxygen therapy - Hemodynamically unstable supply.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-09; Primary Completion 2015-03 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Heart Rate Variability | one hour
  It will be analyzed the uptake of heart rate variability by means of the heart rate monitor Polar ® brand, model RS800CX where FC signal is received by a strap to the signal receiver, to be placed on the thorax at the level of voluntary xiphoid process. This capture is stored in the Polar monitor and transferred to the software Polar ProTrainer program by means of an emission of infrared signals interface, where they are stored and subsequently exported to TXT format, which subsequently can be analyzed by a math routine in Kubios HRV® program. Volunteers will be asked to remain at rest for a period of 10 min, avoiding talking to the researcher so that the heart rate does not undergo changes.
Oxidative stress | one hour
  Morphological evaluation of oxidative stress in the blood plasma is performed by the so called Optical Microscopy Test for In Vitro Analysis Cell or HLB Test. The fingertip of the fourth finger of the previously sanitized hand with alcohol, will collect a drop of blood next to a microscope slide through five light touch of this blade next to the drop .
  At the end of this period, the morphology of this clot is microscopically observed under a 40-fold increase in optical microscope brand Nikon® model Binocular E200 Standard and its qualitative graduation will be recorded by the camera attached Nikon® mark on a spreadsheet to later analysis. The observation of morphological patterns of the different obtained clots will be held in the first image taken on each of the blades and the evaluation will be conducted through the program called OxyScanner® developed and marketed by Aldea Global Soluciones (AGS).

SECONDARY OUTCOMES:
Hospitalization time evaluation | 1 month
  investigate the volunteers of stay in both intervention groups using evaluation of the patients medical records

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Batagello, PHD, Study Director — Universidade Metodista de Piracicaba
Locations (1):
- Hospital de Clínicas Gaspar Viana, Belém, Pará, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The data of the volunteers will be kept confidential , being only used the amount of data for publication in journals with the period until 2017

REFERENCES:
- [Background] Laitio TT, Huikuri HV, Koskenvuo J, Jalonen J, Makikallio TH, Helenius H, Kentala ES, Hartiala J, Scheinin H. Long-term alterations of heart rate dynamics after coronary artery bypass graft surgery. Anesth Analg. 2006 Apr;102(4):1026-31. doi: 10.1213/01.ane.0000198674.90500.59. PMID 16551892
- [Result] Brasher PA, McClelland KH, Denehy L, Story I. Does removal of deep breathing exercises from a physiotherapy program including pre-operative education and early mobilisation after cardiac surgery alter patient outcomes? Aust J Physiother. 2003;49(3):165-73. doi: 10.1016/s0004-9514(14)60236-1. PMID 12952516
- [Result] Burtin C, Clerckx B, Robbeets C, Ferdinande P, Langer D, Troosters T, Hermans G, Decramer M, Gosselink R. Early exercise in critically ill patients enhances short-term functional recovery. Crit Care Med. 2009 Sep;37(9):2499-505. doi: 10.1097/CCM.0b013e3181a38937. PMID 19623052
- [Result] Aubert AE, Seps B, Beckers F. Heart rate variability in athletes. Sports Med. 2003;33(12):889-919. doi: 10.2165/00007256-200333120-00003. PMID 12974657
- [Result] Karemaker JM, Lie KI. Heart rate variability: a telltale of health or disease. Eur Heart J. 2000 Mar;21(6):435-7. doi: 10.1053/euhj.1999.1969. No abstract available. PMID 10681483
- [Result] Sachdev S, Davies KJ. Production, detection, and adaptive responses to free radicals in exercise. Free Radic Biol Med. 2008 Jan 15;44(2):215-23. doi: 10.1016/j.freeradbiomed.2007.07.019. Epub 2007 Jul 31. PMID 18191757
- [Result] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068
- [Result] Truong AD, Fan E, Brower RG, Needham DM. Bench-to-bedside review: mobilizing patients in the intensive care unit--from pathophysiology to clinical trials. Crit Care. 2009;13(4):216. doi: 10.1186/cc7885. Epub 2009 Jul 13. PMID 19664166
- [Result] Silva AP, Maynard K, Cruz MR. Effects of motor physical therapy in critically ill patients: literature review. Rev Bras Ter Intensiva. 2010 Mar;22(1):85-91. English, Portuguese. PMID 25303704
- [Result] Vaishnav S, Stevenson R, Marchant B, Lagi K, Ranjadayalan K, Timmis AD. Relation between heart rate variability early after acute myocardial infarction and long-term mortality. Am J Cardiol. 1994 Apr 1;73(9):653-7. doi: 10.1016/0002-9149(94)90928-8. PMID 8166060
- [Result] Wright DJ, Williams SG, Riley R, Marshall P, Tan LB. Is early, low level, short term exercise cardiac rehabilitation following coronary bypass surgery beneficial? A randomised controlled trial. Heart. 2002 Jul;88(1):83-4. doi: 10.1136/heart.88.1.83. No abstract available. PMID 12067954
- [Result] Zafiropoulos B, Alison JA, McCarren B. Physiological responses to the early mobilisation of the intubated, ventilated abdominal surgery patient. Aust J Physiother. 2004;50(2):95-100. doi: 10.1016/s0004-9514(14)60101-x. PMID 15151493